CLINICAL TRIAL: NCT02706886
Title: A Phase 1/2, Single-Blind, Placebo-Controlled, Single and Multiple Ascending Dose Safety, Tolerability, Pharmacokinetic and Pharmacodynamics Study of Subcutaneously Administered ALN-GO1 in Healthy Adult Subjects, and Patients With Primary Hyperoxaluria Type 1
Brief Title: Study of Lumasiran in Healthy Adults and Patients With Primary Hyperoxaluria Type 1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALN-GO1-001; 2015-004407-23 (EudraCT Number)
Record Dates: First submitted 2016-03-03; First posted 2016-03-11 (Estimated); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Primary Hyperoxaluria Type 1 (PH1)
Keywords: PH1; Primary Hyperoxaluria; RNAi therapeutic; siRNA; AGT
MeSH Terms: conditions — Primary hyperoxaluria type 1; Hyperoxaluria, Primary | interventions — lumasiran

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A: SAD: Placebo (Placebo Comparator): A single dose of matching placebo will be administered subcutaneously (SC).
  Interventions: Drug: Placebo
- Part A: SAD: Lumasiran 0.3 mg/kg (Experimental): A single dose of 0.3 mg/kg lumasiran will be administered SC.
  Interventions: Drug: Lumasiran
- Part A: SAD: Lumasiran 1.0 mg/kg (Experimental): A single dose of 1.0 mg/kg lumasiran will be administered SC.
  Interventions: Drug: Lumasiran
- Part A: SAD: Lumasiran 3.0 mg/kg (Experimental): A single dose of 3.0 mg/kg lumasiran will be administered SC.
  Interventions: Drug: Lumasiran
- Part A: SAD: Lumasiran 6.0 mg/kg (Experimental): A single dose of 6.0 mg/kg lumasiran will be administered SC.
  Interventions: Drug: Lumasiran
- Part B: MAD: Placebo (Placebo Comparator): Participants with primary hyperoxaluria type 1 (PH1) will be treated with placebo matching one of the lumasiran dosages in the lumasiran arms (one placebo participant for each lumasiran arm). At Day 85 these placebo treated participants will cross over to their respective Part B lumasiran arms in the Part B: MAD Study Day 85-End of Study Period and will then be treated with lumasiran. The estimated total time on study was up to 546 days.
  Interventions: Drug: Placebo
- Part B: MAD: Lumasiran 1.0 mg/kg qM (Experimental): Participants with PH1 will be treated with 1.0 mg/kg lumasiran SC once monthly (qM) on Days 1, 29 and 57. The estimated total time on study is up to 546 days. One participant from the Part B: MAD: Placebo arm will cross over to this lumasiran arm at Day 85. For this participant treatment with lumasiran starts at Day 85.
  Interventions: Drug: Lumasiran
- Part B: MAD: Lumasiran 3.0 mg/kg qM (Experimental): Participants with PH1 will be treated with 3.0 mg/kg lumasiran SC qM on Days 1, 29 and 57. The estimated total time on study is up to 546 days. One participant from the Part B: MAD: Placebo arm will cross over to this lumasiran arm at Day 85. For this participant treatment with lumasiran starts at Day 85.
  Interventions: Drug: Lumasiran
- Part B: MAD: Lumasiran 3.0 mg/kg q3M (Experimental): Participants with PH1 will be treated with 3.0 mg/kg lumasiran SC once every three months (q3M) on Days 1 and 85. The estimated total time on study is up to 546 days. One participant from the Part B: MAD: Placebo arm will cross over to this lumasiran arm at Day 85. For this participant treatment with lumasiran starts at Day 85.
  Interventions: Drug: Lumasiran

INTERVENTIONS:
Drug: Lumasiran — Lumasiran will be administered SC once in Part A. In Part B lumasiran will be administered SC qM (Days 1, 29 and 57) or q3M (Days 1 and 85).
  Other Names: ALN-GO1
  Arms: Part A: SAD: Lumasiran 0.3 mg/kg; Part A: SAD: Lumasiran 1.0 mg/kg; Part A: SAD: Lumasiran 3.0 mg/kg; Part A: SAD: Lumasiran 6.0 mg/kg; Part B: MAD: Lumasiran 1.0 mg/kg qM; Part B: MAD: Lumasiran 3.0 mg/kg q3M; Part B: MAD: Lumasiran 3.0 mg/kg qM
Drug: Placebo — Matching placebo (sterile saline: 0.9% sodium chloride [NaCl]) will be administered SC once in Part A. In Part B matching placebo will be administered SC qM (Days 1, 29 and 57) or q3M (Days 1 and 85).
  Arms: Part A: SAD: Placebo; Part B: MAD: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single-ascending doses (SAD) and multiple-ascending doses (MAD) of lumasiran in healthy adult volunteers and subjects with primary hyperoxaluria type 1 (PH1). In Part A, single ascending dose (SAD) part, healthy adults were dosed with lumasiran or placebo once. In Part B, multiple ascending doses (MAD) part, patients with primary hyperoxaluria type 1 (PH1) were dosed with lumasiran or placebo. All patients that initially received placebo received lumasiran after completing placebo dosing.

ELIGIBILITY:
Inclusion Criteria for Parts A and B:

* Women of child bearing potential must have a negative pregnancy test, cannot be breastfeeding, and must be willing to use contraception.
* Willing to provide written informed consent and to comply with study requirements.

Additional Inclusion Criteria for Part B:

* Confirmation of PH1 disease
* Meet 24 hour urine oxalate excretion requirements
* Estimated glomerular filtration rate (GFR) of >45 mL/min/1.73m^2
* If taking Vitamin B6 (pyridoxine), must have been on stable regimen for at least 90 days

Exclusion Criteria for Parts A and B:

* Clinically significant health concerns (with the exception of PH1 for patients in Part B)
* Clinically significant electrocardiogram (ECG) abnormalities
* Abnormal for aspartate aminotransferase (AST)/alanine aminotransferase (ALT) and any other clinical safety laboratory result considered clinically significant
* Received an investigational agent within 3 months before the first dose of study drug or are in follow-up of another clinical study
* Known history of allergic reaction to an oligonucleotide or N-acetylgalactosamine (GalNAc)
* History of intolerance to subcutaneous injection

Ages: 6 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy McGregor, MD, MSCI, Study Director — Alnylam Pharmaceuticals
Locations (9):
- France (3):
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Lyon
  - Clinical Trial Site, Paris
- Clinical Trial Site, Bonn, Germany
- Israel (2):
  - Clinical Trial Site, Haifa
  - Clinical Trial Site, Jerusalem
- Clinical Trial Site, Amsterdam, Netherlands
- United Kingdom (2):
  - Clinical Trial Site, Birmingham
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Badri P, Kolachana K, Duong A, Lasko M, Nandi T, Mehrotra N, Robbie GJ. Platform Assessment of Concentration-QTc Relationship Across GalNAc-siRNA Molecules. Clin Pharmacokinet. 2025 Dec 12. doi: 10.1007/s40262-025-01606-0. Online ahead of print. PMID 41388232
- [Derived] Frishberg Y, Deschenes G, Groothoff JW, Hulton SA, Magen D, Harambat J, Van't Hoff WG, Lorch U, Milliner DS, Lieske JC, Haslett P, Garg PP, Vaishnaw AK, Talamudupula S, Lu J, Habtemariam BA, Erbe DV, McGregor TL, Cochat P; study collaborators. Phase 1/2 Study of Lumasiran for Treatment of Primary Hyperoxaluria Type 1: A Placebo-Controlled Randomized Clinical Trial. Clin J Am Soc Nephrol. 2021 Jul;16(7):1025-1036. doi: 10.2215/CJN.14730920. Epub 2021 May 13. PMID 33985991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at ten sites in Germany, France, the United Kingdom, Israel, and the Netherlands.
Pre-assignment Details: In Part A, single ascending dose (SAD) part, healthy adults were dosed with lumasiran or placebo once. In Part B, multiple ascending doses (MAD) part, patients with primary hyperoxaluria type 1 (PH1) were dosed with lumasiran or placebo. All patients, who initially received placebo, received lumasiran after completing placebo dosing.
Groups:
- Part A: SAD: Placebo: A single dose of matching placebo was administered subcutaneously (SC).
- Part A: SAD: Lumasiran 0.3 mg/kg: A single dose of 0.3 mg/kg lumasiran was administered SC.
- Part A: SAD: Lumasiran 1.0 mg/kg: A single dose of 1.0 mg/kg lumasiran was administered SC.
- Part A: SAD: Lumasiran 3.0 mg/kg: A single dose of 3.0 mg/kg lumasiran was administered SC.
- Part A: SAD: Lumasiran 6.0 mg/kg: A single dose of 6.0 mg/kg lumasiran was administered SC.
- Part B: MAD: Placebo: Participants with primary hyperoxaluria type 1 (PH1) were treated with placebo matching one of the lumasiran dosages in the lumasiran arms (one placebo participant for each lumasiran arm). At Day 85 these placebo-treated participants crossed over to their respective Part B lumasiran arms in Part B: MAD Study Day 85-End of Study and were then treated with lumasiran. The estimated total time on study was up to 546 days.
- Part B: MAD: Lumasiran 1.0 mg/kg qM: Participants with PH1 were treated with 1.0 mg/kg lumasiran SC once monthly (qM) on Days 1, 29 and 57. The estimated total time on study was up to 546 days. One participant from the Part B: MAD: Placebo arm crossed over to this lumasiran arm at Day 85. For this participant treatment with lumasiran started at Day 85.
- Part B: MAD: Lumasiran 3.0 mg/kg qM: Participants with PH1 were treated with 3.0 mg/kg lumasiran SC qM on Days 1, 29 and 57. The estimated total time on study was up to 546 days. One participant from the Part B: MAD: Placebo arm crossed over to this lumasiran arm at Day 85. For this participant treatment with lumasiran started at Day 85.
- Part B: MAD: Lumasiran 3.0 mg/kg q3M: Participants with PH1 were treated with 3.0 mg/kg lumasiran SC once every three months (q3M) on Days 1 and 85. The estimated total time on study was up to 546 days. One participant from the Part B: MAD: Placebo arm crossed over to this lumasiran arm at Day 85. For this participant treatment with lumasiran started at Day 85.
Period: Part A: SAD Period
Arm/Group | Part A: SAD: Placebo | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Started | 8 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
Completed | 8 | 6 | 6 | 4 | 6 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Period: Part B: MAD Study Days 1-85
Arm/Group | Part A: SAD: Placebo | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Started | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 7 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 7 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: MAD Study Day 85-End of Study
Arm/Group | Part A: SAD: Placebo | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Started | 0 | 0 | 0 | 0 | 0 | 0 | 8 (One participant from the Part B: MAD: Placebo arm crossed over to this lumasiran arm.) | 8 (One participant from the Part B: MAD: Placebo arm crossed over to this lumasiran arm.) | 4 (One participant from the Part B: MAD: Placebo arm crossed over to this lumasiran arm.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set consisted of all healthy participants and participants who received at least 1 dose of study drug (lumasiran, placebo), grouped according to actual treatment received during the first period that they entered the study.
Groups:
- Part A: SAD: Placebo: A single dose of matching placebo was administered SC.
- Total: Total of all reporting groups
Arm/Group | Part A: SAD: Placebo | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 3 | 7 | 7 | 3 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (6.25) | 28.8 (7.36) | 30.2 (7.81) | 27.3 (3.44) | 28.8 (5.46) | 20.7 (19.40) | 14.0 (9.93) | 15.4 (7.89) | 9.7 (5.51) | 23.6 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 3 | 3 | 5 | 1 | 6 | 4 | 2 | 29
  Male | 3 | 6 | 3 | 3 | 1 | 2 | 1 | 3 | 1 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 7 | 5 | 6 | 6 | 5 | 3 | 7 | 7 | 3 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  White | 7 | 6 | 5 | 3 | 4 | 2 | 5 | 5 | 3 | 40
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigational subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
Time Frame: Part A (SAD): Up to 405 days; Part B (MAD): Up to 546 days
Population: Safety Analysis Set consisted of all healthy participants and patients, who received at least 1 dose of study drug (lumasiran, placebo), grouped according to actual treatment received. Part B participants who crossed over from placebo to the lumasiran arms are included in the placebo arm as well as lumasiran arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SAD: Placebo | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 3 | 8 | 8 | 4
Participants | 5 | 6 | 2 | 6 | 6 | 2 | 8 | 7 | 4

2. Secondary Outcome: Maximum Concentration (Cmax) of Lumasiran in Plasma
Description: Samples for Part A were collected only on Day 1; Part B on Days 1 and 57 for qM and on Days 1 and 85 for q3M arm groups.
Time Frame: Part A (SAD): Day 1: predose, 30 minutes (min), 1 hour (h), 2 h, 4 h, 6 h, 8 h and 24 h; Part B (MAD): Days 1 and 57 for qM dosing and Days 1 and 85 for q3M dosing: predose, 30 min, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h and 48 h
Population: Pharmacokinetic (PK) Analysis Set consisted of all healthy participants and patients who received at least 1 dose of lumasiran and had at least 1 postdose sample for PK parameters and who had evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 4
ng/mL
  Day 1 | 39.7940 (8.58882) | 204.3748 (111.68091) | 533.4527 (160.11060) | 1176.1302 (199.89797) | 324.1386 (489.71104) | 582.4515 (266.90105) | 432.2798 (245.02660)
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8 | 0
  Day 57 |  |  |  |  | 147.6780 (67.97968) | 701.1708 (511.63001) |
  Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Day 85 |  |  |  |  |  |  | 411.5613 (174.92146)

3. Secondary Outcome: Time to Cmax (Tmax) of Lumasiran in Plasma
Description: Samples for Part A were collected only on Day 1; Part B on Days 1 and 57 for qM and on Days 1 and 85 for q3M arm groups.
Time Frame: Part A (SAD): Day 1: predose, 30 min, 1 h, 2 h, 4 h, 6 h, 8 h and 24 h; Part B (MAD): Days 1 and 57 for qM dosing and Days 1 and 85 for q3M dosing: predose, 30 min, 1 h, 2 h, 4 h, 6 h, 8 h, 12 h, 24 h and 48 h
Population: PK Analysis Set consisted of all healthy participants and patients who received at least 1 dose of lumasiran and had at least 1 postdose sample for PK parameters and who had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 4
hours
  Day 1 | 5.0167 [4.000 to 8.017] | 1.5000 [0.517 to 8.000] | 3.0000 [0.500 to 8.000] | 7.0000 [0.500 to 8.067] | 3.9917 [0.567 to 5.967] | 4.9917 [0.533 to 12.000] | 9.0000 [5.783 to 12.017]
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8 | 0
  Day 57 |  |  |  |  | 3.0417 [0.500 to 6.000] | 2.9833 [0.500 to 8.000] |
  Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Day 85 |  |  |  |  |  |  | 5.9833 [4.050 to 7.950]

4. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Time of Last Measurable Concentration (AUC0-last) of Lumasiran in Plasma
Description: Samples for Part A were collected only on Day 1; Part B on Days 1 and 57 for qM and on Days 1 and 85 for q3M arm groups.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- Part A: SAD: Lumasiran 0.3 mg/kg: A single dose of 0.3 mg/kg lumasiran was administered subcutaneously (SC).
Arm/Group | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 8 | 4
h*ng/mL
  Day 1 | 293.5232 (96.86989) | 1899.8119 (558.25326) | 7211.5890 (1125.64173) | 16778.0579 (4380.15325) | 1428.0412 (697.85233) | 7400.2181 (2331.89843) | 6337.9082 (3840.03340)
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 8 | 0
  Day 57 |  |  |  |  | 1608.1457 (708.95156) | 7959.7873 (1726.57675) |
  Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Day 85 |  |  |  |  |  |  | 5136.3462 (2757.90139)

5. Secondary Outcome: Terminal Half-life (t1/2) of Lumasiran in Plasma
Description: Samples for Part A were collected only on Day 1; Part B on Days 1 and 57 for qM and on Days 1 and 85 for q3M arm groups.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 2 | 2 | 1 | 4 | 5 | 1
hours
  Day 1 | 7.0655 (0.37379) | 5.9798 (1.52471) | 3.4683 (NA) — SD was not calculated for arms with data for 1 participant. | 3.2670 (1.52759) | 5.4574 (3.49432) | 7.8028 (NA) — SD was not calculated for arms with data for 1 participant.
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 4 | 4 | 0
  Day 57 |  |  |  | 7.8090 (4.52009) | 5.8356 (3.12156) |
  Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1
  Day 85 |  |  |  |  |  | 4.6694 (NA) — SD was not calculated for arms with data for 1 participant.

6. Secondary Outcome: Fraction Excreted in Urine in 24 Hours (Fe0-24) of Lumasiran
Description: Samples for Part A were collected only on Day 1; Part B on Days 1 and 57 for qM and on Days 1 and 85 for q3M arm groups.
Time Frame: Part A (SAD): Day 1: pooled urine 0-4 h, 4-8 h and 8-24 h; Part B (MAD): Part B (MAD phase): Days 1 and 57 for qM dosing and Days 1 and 85 for q3M dosing: pooled urine 0-4 h, 4-8 h, 8-12 h and 12-24 h
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage fractional excretion
Arm/Group | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 8 | 7 | 4
percentage fractional excretion
  Day 1: number analyzed (Participants) | 6 | 6 | 6 | 5 | 7 | 7 | 4
  Day 1 | 17.4219 (2.44129) | 19.0713 (3.88914) | 21.0472 (5.36667) | 25.7931 (3.25937) | 11.0895 (3.74207) | 11.1877 (6.07719) | 7.1691 (2.37465)
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 6 | 0
  Day 57 |  |  |  |  | 9.4698 (4.21949) | 12.4604 (4.02897) |
  Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Day 85 |  |  |  |  |  |  | 13.6938 (3.60004)

7. Secondary Outcome: Renal Clearance (CLR) of Lumasiran
Description: Samples for Part A were collected only on Day 1; Part B on Days 1 and 57 for qM and on Days 1 and 85 for q3M arm groups.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 1 | 5 | 6 | 5 | 7 | 6 | 4
L/h
  Day 1: number analyzed (Participants) | 1 | 5 | 6 | 5 | 6 | 6 | 4
  Day 1 | 8.7817 (NA) — SD was not calculated for arms with data for 1 participant. | 5.4906 (2.07402) | 5.8211 (1.31377) | 6.3417 (1.15497) | 2.2612 (1.17616) | 2.3818 (1.13067) | 2.0564 (1.20600)
  Day 57: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 6 | 0
  Day 57 |  |  |  |  | 1.9610 (1.11228) | 2.5150 (0.80386) |
  Day 85: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Day 85 |  |  |  |  |  |  | 3.3663 (1.18371)

8. Secondary Outcome: Baseline Plasma Glycolate Concentration
Description: The pharmacodynamic (PD) outcome measure of plasma glycolate concentration could only be calculated for Part A. Due to an issue with the plasma glycolate assay at the testing laboratory the data for Part B could not be calculated.
Time Frame: Part A (SAD): Baseline, Part B (MAD): Baseline
Population: PD Analysis Set consisted of all participants who received at least 1 dose of study drug (lumasiran, placebo) and had at least 1 postdose blood sample available that was evaluable for PD assessments. Due to an issue with plasma glycolate assay at the testing laboratory the data for Part B could not be calculated.
Measure: Mean (Standard Deviation); unit: umol/L
Groups:
- Part B: MAD: Placebo: Participants with primary hyperoxaluria type 1 (PH1) were treated with placebo matching one of the lumasiran dosages in the lumasiran arms (one placebo participant for each lumasiran arm). At Day 85 these placebotreated participants crossed over to their respective Part B lumasiran arms in Part B: MAD Study Day 85-End of Study and were then treated with lumasiran. The estimated total time on study was up to 546 days.
Arm/Group | Part A: SAD: Placebo | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
umol/L | 5.1 (1.73) | 5.3 (1.51) | 5.7 (1.97) | 6.2 (2.56) | 4.8 (1.72) |  |  |  |

9. Secondary Outcome: Percentage Change From Baseline in Plasma Glycolate Concentration
Description: The PD outcome measure of plasma glycolate concentration could only be calculated for Part A. Due to an issue with the plasma glycolate assay at the testing laboratory the data for Part B could not be calculated.
Time Frame: Part A (SAD): Days 15, 29, 57 and 85; Part B (MAD): Days 15, 29, 57, 85
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Part A: SAD: Placebo | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 0 | 0 | 0 | 0
percentage change from baseline
  Day 15 | 18.3 (67.19) | 58.3 (55.29) | 48.5 (82.99) | 56.4 (28.50) | 59.5 (49.00) |  |  |  |
  Day 29 | 22.4 (46.83) | 32.9 (57.67) | 70.6 (82.74) | 146.4 (81.99) | 390.1 (270.40) |  |  |  |
  Day 57 | 126.7 (242.68) | 66.3 (38.07) | 109.8 (124.29) | 230.1 (180.36) | 730.4 (439.54) |  |  |  |
  Day 85: number analyzed (Participants) | 8 | 6 | 6 | 5 | 6 | 0 | 0 | 0 | 0
  Day 85 | 31.2 (131.04) | 15.6 (100.54) | 40.7 (110.75) | 196.2 (152.41) | 731.3 (375.02) |  |  |  |

10. Secondary Outcome: Baseline Spot Urine Glycolate:Creatinine Ratio in Part A
Description: The endpoint was only measured in Part A.
Time Frame: Part A (SAD): Baseline
Population: PD Analysis Set for Part A consisted of all healthy participants who received at least 1 dose of study drug (lumasiran, placebo) and had at least 1 postdose blood and/or urine sample available that was evaluable for PD assessments.
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Part A: SAD: Placebo | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
mg/g | 12.4 (4.63) | 15.7 (4.27) | 15.7 (3.14) | 13.0 (3.52) | 14.8 (4.31)

11. Secondary Outcome: Percentage Change From Baseline in Spot Urine Glycolate:Creatinine Ratio in Part A
Description: The endpoint was only measured in Part A.
Time Frame: Part A (SAD): Days 29 and 57
Population: PD Analysis Set in Part A consisted of all healthy participants who received at least 1 dose of study drug (lumasiran, placebo) and had at least 1 postdose blood and/or urine sample available that was evaluable for PD assessments.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Part A: SAD: Placebo | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
percentage change from baseline
  Day 29 | 8.1 (43.42) | 32.5 (22.6) | 82.9 (65.00) | 109.1 (66.51) | 210.5 (199.30)
  Day 57 | 73.8 (108.9) | 38.0 (50.62) | 47.8 (41.03) | 215.0 (178.72) | 310.7 (94.51)

12. Secondary Outcome: Baseline of 24 Hour Urine Oxalate Corrected for BSA in Part B
Description: The endpoint was only measured in Part B.
Time Frame: Part B (MAD): Baseline
Population: PD Analysis Set in Part B consisted of all patients with PH1 who received at least 1 dose of study drug (lumasiran, placebo) and had at least 1 postdose blood and/or urine sample available that was evaluable for PD assessments.
Measure: Mean (Standard Deviation); unit: mmol/24h/1.73m^2
Arm/Group | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 3 | 8 | 8 | 4
mmol/24h/1.73m^2 | 1.96 (0.321) | 1.73 (0.696) | 1.84 (0.621) | 1.30 (0.350)

13. Secondary Outcome: Percentage Change From Baseline of 24 Hour Urine Oxalate Corrected for BSA in Part B
Description: The endpoint was only measured in Part B.
Time Frame: Part B (MAD): 24 hour urine collections on Days 29, 57, 85, 113, 141, 169, 197
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 2 | 8 | 8 | 4
percentage change from baseline
  Day 29: number analyzed (Participants) | 1 | 7 | 7 | 4
  Day 29 | -2.4 (NA) — SD was not calculated for arms with data for 1 participant. | -41.1 (24.76) | -57.5 (10.84) | -49.2 (5.40)
  Day 57: number analyzed (Participants) | 2 | 7 | 8 | 4
  Day 57 | -27.8 (47.11) | -49.7 (20.08) | -72.5 (10.70) | -49.1 (5.82)
  Day 85: number analyzed (Participants) | 1 | 8 | 7 | 3
  Day 85 | 9.1 (NA) — SD was not calculated for arms with data for 1 participant. | -65.6 (16.64) | -68.4 (10.60) | -53.3 (3.66)
  Day 113: number analyzed (Participants) | 0 | 7 | 6 | 4
  Day 113 |  | -61.4 (12.24) | -78.1 (7.80) | -59.1 (20.75)
  Day 141: number analyzed (Participants) | 0 | 7 | 7 | 2
  Day 141 |  | -64.6 (13.55) | -73.5 (8.11) | -68.4 (3.21)
  Day 169: number analyzed (Participants) | 0 | 8 | 7 | 3
  Day 169 |  | -61.6 (14.19) | -69.3 (9.61) | -48.7 (14.19)
  Day 197: number analyzed (Participants) | 0 | 6 | 7 | 4
  Day 197 |  | -63.8 (13.85) | -71.2 (11.70) | -52.7 (6.38)

14. Secondary Outcome: Baseline 24 Hour Urine Glycolate:Creatinine Ratio in Part B - Initial 85 Days
Description: The endpoint was only measured during the initial 85 days in Part B.
Time Frame: Part B (MAD): Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 3 | 7 | 7 | 3
mg/g | 193 (117.2) | 241 (85.6) | 289 (146.0) | 281 (139.0)

15. Secondary Outcome: Percentage Change From Baseline of 24 Hour Urine Glycolate:Creatinine Ratio in Part B - Initial 85 Days
Description: The endpoint was only measured during the initial 85 days in Part B.
Time Frame: Part B (MAD): 24 hour urine collections on Days 29, 57 and 85
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 3 | 7 | 7 | 3
percentage change from baseline
  Day 29 | -15.1 (6.47) | 53.1 (42.18) | 31.4 (35.99) | 33.0 (36.37)
  Day 57 | -13.8 (29.02) | 82.3 (40.12) | 42.3 (57.56) | 81.8 (35.66)
  Day 85: number analyzed (Participants) | 3 | 7 | 7 | 2
  Day 85 | -23.0 (10.45) | 71.0 (55.62) | 43.7 (62.15) | 42.0 (20.86)

16. Secondary Outcome: Baseline Creatinine Clearance Corrected for BSA in Part B
Time Frame: Part B (MAD): Baseline
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 3 | 8 | 8 | 4
mL/min/1.73 m^2 | 64.389 (19.8024) | 108.149 (44.1783) | 86.268 (22.1226) | 88.251 (30.0118)

17. Secondary Outcome: Percentage Change From Baseline of Creatinine Clearance Corrected for BSA in Part B
Time Frame: Part B (MAD): Days 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337, 365, 393, 421, 449
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
Number analyzed (Participants) | 2 | 8 | 8 | 4
percentage change from baseline
  Day 29: number analyzed (Participants) | 1 | 7 | 7 | 4
  Day 29 | 9.019 (NA) — Standard Deviation is not calculated for arms with one participant | -6.672 (11.9614) | -0.624 (15.1771) | 2.748 (5.6858)
  Day 57: number analyzed (Participants) | 2 | 7 | 8 | 4
  Day 57 | 20.184 (23.5572) | -8.426 (19.7271) | 4.505 (35.2457) | 37.030 (56.1210)
  Day 85: number analyzed (Participants) | 1 | 8 | 7 | 2
  Day 85 | -5.945 (NA) — Standard Deviation is not calculated for arms with one participant | -13.536 (22.8679) | -3.720 (22.6231) | -6.113 (43.5441)
  Day 113: number analyzed (Participants) | 0 | 7 | 6 | 4
  Day 113 |  | -14.424 (24.1107) | 3.444 (29.6749) | 7.570 (40.5928)
  Day 141: number analyzed (Participants) | 0 | 7 | 7 | 2
  Day 141 |  | -8.804 (27.4802) | 9.315 (27.5044) | -30.691 (12.8912)
  Day 169: number analyzed (Participants) | 0 | 8 | 7 | 1
  Day 169 |  | -19.796 (31.7492) | -8.544 (14.8481) | 20.210 (NA) — Standard Deviation is not calculated for arms with one participant
  Day 197: number analyzed (Participants) | 0 | 6 | 7 | 4
  Day 197 |  | -8.546 (13.5672) | -13.513 (25.0560) | 28.857 (22.1891)
  Day 225: number analyzed (Participants) | 0 | 6 | 8 | 3
  Day 225 |  | -18.221 (14.2322) | 29.013 (53.5563) | -14.964 (9.9130)
  Day 253: number analyzed (Participants) | 0 | 6 | 7 | 0
  Day 253 |  | -5.140 (19.2839) | 10.232 (24.4929) |
  Day 281: number analyzed (Participants) | 0 | 6 | 6 | 0
  Day 281 |  | -14.283 (22.6126) | 5.841 (13.0381) |
  Day 309: number analyzed (Participants) | 0 | 5 | 4 | 0
  Day 309 |  | -0.403 (34.6839) | 8.441 (11.5329) |
  Day 337: number analyzed (Participants) | 0 | 4 | 4 | 0
  Day 337 |  | -5.168 (31.0756) | 8.688 (24.2094) |
  Day 365: number analyzed (Participants) | 0 | 2 | 2 | 0
  Day 365 |  | 2.268 (33.7565) | 9.201 (14.4856) |
  Day 393: number analyzed (Participants) | 0 | 3 | 2 | 0
  Day 393 |  | -11.942 (45.3027) | -4.484 (12.6320) |
  Day 421: number analyzed (Participants) | 0 | 3 | 2 | 0
  Day 421 |  | 7.610 (11.2195) | -6.498 (12.9022) |
  Day 449: number analyzed (Participants) | 0 | 0 | 2 | 0
  Day 449 |  |  | -15.093 (10.3705) |

ADVERSE EVENTS:
Time Frame: Part A (SAD phase): Up to 405 days; Part B (MAD phase): Up to 546 days
Description: Safety Analysis Set consisted of all healthy participants and patients who received at least 1 dose of study drug (lumasiran, placebo), grouped according to actual treatment received. Part B participants who crossed over from placebo to the lumasiran arms are included in the placebo arm as well as lumasiran arms and adverse events are reported based on the treatment received at the time of the event.
Groups:
- Part A: SAD: Placebo: A single dose of matching placebo was administered.
- Part B: MAD: Placebo: Participants with primary hyperoxaluria type 1 (PH1) were treated with placebo matching one of the lumasiran dosages in the lumasiran arms (one placebo participant for each lumasiran arm). At Day 85 these placebo-treated participants crossed over to their respective Part B lumasiran arms in the All-Lumasiran-Treated Period. The estimated total time on study was up to 546 days.
- Part B: MAD: Lumasiran 1.0 mg/kg qM: Participants with PH1 were treated with 1.0 mg/kg lumasiran SC once monthly (qM) on Days 1, 29 and 57. The estimated total time on study was up to 546 days.
- Part B: MAD: Lumasiran 3.0 mg/kg qM: Participants with PH1 were treated with 3.0 mg/kg lumasiran SC qM on Days 1, 29 and 57. The estimated total time on study was up to 546 days.
- Part B: MAD: Lumasiran 3.0 mg/kg q3M: Participants with PH1 were treated with 3.0 mg/kg lumasiran SC once every three months (q3M) on Days 1 and 85. The estimated total time on study was up to 546 days.
Arm/Group | Part A: SAD: Placebo | Part A: SAD: Lumasiran 0.3 mg/kg | Part A: SAD: Lumasiran 1.0 mg/kg | Part A: SAD: Lumasiran 3.0 mg/kg | Part A: SAD: Lumasiran 6.0 mg/kg | Part B: MAD: Placebo | Part B: MAD: Lumasiran 1.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg qM | Part B: MAD: Lumasiran 3.0 mg/kg q3M
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/8 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 1/3 | 1/8 | 3/8 | 0/4
Other Adverse Events (participants affected / at risk) | 5/8 | 6/6 | 3/6 | 6/6 | 6/6 | 2/3 | 7/8 | 7/8 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SAD: Placebo (N=8) | Part A: SAD: Lumasiran 0.3 mg/kg (N=6) | Part A: SAD: Lumasiran 1.0 mg/kg (N=6) | Part A: SAD: Lumasiran 3.0 mg/kg (N=6) | Part A: SAD: Lumasiran 6.0 mg/kg (N=6) | Part B: MAD: Placebo (N=3) | Part B: MAD: Lumasiran 1.0 mg/kg qM (N=8) | Part B: MAD: Lumasiran 3.0 mg/kg qM (N=8) | Part B: MAD: Lumasiran 3.0 mg/kg q3M (N=4)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SAD: Placebo (N=8) | Part A: SAD: Lumasiran 0.3 mg/kg (N=6) | Part A: SAD: Lumasiran 1.0 mg/kg (N=6) | Part A: SAD: Lumasiran 3.0 mg/kg (N=6) | Part A: SAD: Lumasiran 6.0 mg/kg (N=6) | Part B: MAD: Placebo (N=3) | Part B: MAD: Lumasiran 1.0 mg/kg qM (N=8) | Part B: MAD: Lumasiran 3.0 mg/kg qM (N=8) | Part B: MAD: Lumasiran 3.0 mg/kg q3M (N=4)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 1 | 4 | 4 | 0 | 0 | 0 | 2
Periodontitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 1 | 3 | 0 | 2 | 2 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Alcoholic hangover (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Caffeine consumption (Social circumstances) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Teething (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site discolouration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Overweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT02706886/SAP_000.pdf
  • Study Protocol (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT02706886/Prot_001.pdf